CLINICAL TRIAL: NCT01022216
Title: A Randomized, Controlled Trial of the Procellera™ Wound Dressing Used With Negative Pressure Wound Therapy (NPWT) in the Healing of Diabetic and Pressure Ulcers of the Foot
Brief Title: Efficacy Study of a Bioelectric Dressing Used With Negative Pressure Wound Therapy to Treat Diabetic and Pressure Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vomaris Innovations (Industry)
Responsible Party: Ronald Guberman, DPM, Director, Podiatric Medical Education, Wyckoff Heights Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XSMP-013
Record Dates: First submitted 2009-11-24; First posted 2009-12-01 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Wound Healing
Keywords: Wound; Skin lesion; Antimicrobial; Bioelectric; Diabetic foot; Pressure Ulcer
MeSH Terms: conditions — Wounds and Injuries; Diabetic Foot; Pressure Ulcer | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- V.A.C.® Therapy (Active Comparator): Vacuum Assisted Closure device that utilizes controlled negative pressure
  Interventions: Device: V.A.C.® Therapy
- Procellera™ Wound Dressing with V.A.C.® Therapy (Experimental): Procellera wound dressing used as a primary contact layer on the wound bed, used in conjunction with NPWT
  Interventions: Device: Procellera™ Wound Dressing with V.A.C.® Therapy

INTERVENTIONS:
Device: Procellera™ Wound Dressing with V.A.C.® Therapy — Dressing indicated for partial and full-thickness wounds. Weekly dressing changes, more frequently if needed. Used as a primary contact layer in conjunction with NPWT.
  Other Names: PROCELLERA™, PROSIT™, Bioelectric
  Arms: Procellera™ Wound Dressing with V.A.C.® Therapy
Device: V.A.C.® Therapy — Vacuum Assisted Closure device that uses controlled negative pressure, with dressing changes 1x/week.
  Other Names: Negative Pressure Wound Therapy, Vacuum Assisted Closure, V.A.C.® Therapy,
  Arms: V.A.C.® Therapy

SUMMARY:
The purpose of this study is to determine whether a bioelectric wound dressing, used in conjunction with Negative Pressure Wound Therapy (NPWT), is effective in the treatment of diabetic and pressure ulcers of the foot.

ELIGIBILITY:
Inclusion Criteria:

* Wound size greater than 1x1 cm
* Wounds must be ≥5 cm away from all other wounds
* Wound size must not be diminished in size greater than 10% between enrollment in study and the prescreening
* Participant must be candidate for negative pressure wound therapy
* Participant agrees to participate in follow-up evaluations
* Participant must be able to read and understand informed consent, and sign the informed consent

Exclusion Criteria:

* Concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study
* Participant is to receive another topical agent (antimicrobials, enzymes, etc.) other than the study dressing (granufoam)
* Participant is to receive Silver granufoam for their wound
* Participant with sensitivity or adverse reactions to silver or zinc
* Pregnancy or nursing an infant or child
* Immunosuppression
* Active or systemic infection
* Participant undergoing active cancer chemotherapy
* Chronic steroid use

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Wound healing over time | 3 months after enrollment

SECONDARY OUTCOMES:
Pain reduction | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Guberman, DPM, Principal Investigator — Wyckoff Heights Medical Center
Locations (1):
- Wyckoff Heights Medical Center, Brooklyn, New York, United States